CLINICAL TRIAL: NCT03803046
Title: Cognitive Impact of Benzodiazepin Withdrawn After Curative Epilepsy Surgery in Children With Focal Epilepsy
Acronym: COGNIBENZO
Status: Terminated | Type: Observational
Why Stopped: Consequences of failing to include.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P160945J; 2017-003685-27 (EudraCT Number)
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Cognitive Impact of Antiepileptic Drugs
Keywords: Benzodiazepin; Children; Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epilepsy is a frequent group of diseases, affecting 1% of the general population with a higher incidence in children. Anti-epileptic drugs are used as part of the drug treatment. Even if children with epilepsy have its own characteristics, as in adults, the choice of an anti-epileptic treatment is also based on the benefit-risk balance. The purpose of the treatment should not only be the seizure control. The occurence of side effects is a major factor to be taken into account. In the special populatIon of children with resistant epilepsy (20 to 30% of epilepsy), the treatment goal is not any more to be seizure free but to achieve the lowest possible frequency of seizures with the lowest level of side effects.

When assessing the benefit-risk balance of antiepileptic treatment, it is important to keep in mind that the child is a developing human being whose main activity is learning. Special attention should be paid to minimize treatments with excessive cognitive consequences. Be particularly wary of combination therapies (combinations of several antiepileptic treatments). Indeed, it is well established that they are more harmful than monotherapy. It is also important to avoid the use of drugs with too strong a cognitive effect. Some molecules such as phenobarbital or topiramate have been the subject of a few studies that have established their deleterious effect on the cognitive level. Among antiepileptics, benzodiazepines are sometimes used as disease-modifying therapy. In France, clobazam is the clonazepam have a Marketing Authorization for children.

However, there is no study to determine whether these molecules have cognitive consequences. In order to have more data to better establish the risk-benefit balance of benzodiazepines in the treatment of children with epilepsy, the investigators wish to conduct work to evaluate the cognitive consequences of benzodiazepines in children treated for epilepsy.

DETAILED DESCRIPTION:
1. Research Assumptions Epilepsy is a frequent group of diseases, affecting 1% of the general population with a higher incidence in children. Anti-epileptic drugs are used as the main treatment. The choice of an anti-epileptic treatment is based on the benefit-risk balance. The purpose of the treatment should not only be efficacy, the presence of side effects is a major factor to be taken into account. Thus, in children with resistant epilepsy (20 to 30% of epilepsy), the objective is not necessarily to be seizure free but to achieve the lowest possible frequency of seizures with the lowest possible side effects.

   When assessing the benefit-risk ratio of antiepileptic treatment, it is important to keep in mind that the child has a developing brain whose main activity is learning. Special attention should be paid to minimize treatment related cognitive consequences. Be particularly wary of combination therapies (combinations of several antiepileptic treatments). Indeed, it is well established that they are more harmful than monotherapy. It is also important to avoid the use of drugs with too strong cognitive effect of their own. Some molecules such as phenobarbital or topiramate have been the subject of a few studies that have established their deleterious effect on the cognitive level. Benzodiazepines are available drug used as antiepileptic drugs. In France, clobazam and clonazepam have a Marketing Authorization for children.

   Although effective in children with epilepsy, benzodiazepines seem to raised a significant number of problems. One of them is the absence of study determining whether these molecules have cognitive consequences. In order to have more data to better establish the risk-benefit balance of benzodiazepines in the treatment of children with epilepsy, the investigators wish to conduct work to evaluate the cognitive consequences of benzodiazepines in children treated for epilepsy.

   Hypothesis tested: Benzodiazepines have cognitive consequences in children treated for epilepsy The investigators will conduct a prospective study on the cognitive impact of benzodiazepine withdrawal after successful curative epilepsy surgery in children. The investigators will focus, through neuropsychological tests, on the working memory and attention abilities of children with drug-resistant epilepsy who require surgery and are receiving a benzodiazepine. The three assessments (pre-surgical (seizures and benzodiazepine); post-surgical (no seizure and benzodiazepine) and post benzodiazepine discontinuation (no seizure and benzodiazepine)) will assess the impact of benzodiazepines on working memory and attention abilities.

   The data from this study will allow physicians to better understand the balance of benefit and risk balance of benzodiazepine use in children with epilepsy. These data could lead to the writing of a good use for the treatment of epilepsy in children and avoid misuse if the cognitive impact is significant.
2. Description of the studied population and justification for its choice Children followed for drug-resistant epilepsy in preoperative assessment will be selected by the coordinator's team or one of the partners. Indeed, only this methodology (pre- and post-operative comparison with and without benzodiazepine) will make it possible to answer the question asked and in particular the comparison of post-operative evaluation with benzodiazepines with post-operative evaluation after stopping benzodiazepines
3. Benzodiazepin as antiepileptic drugs Efficiency profile: The efficacy spectrum of clobazam and clonazepam is quite broad since these molecules have shown their efficacy in controlled trials on absences, myoclonias, atonic seizures and focal seizures as well as in open trials on generalized tonic-clonic and focal seizures. Some authors have even suggested that clonazepam may be the third line treatment in Lennox-Gastaut syndrome.

   Cognitive side effects: As mentioned above, the cognitive effects of antiepileptics are an important concern in children with epilepsy. This is one of the main point in the benefit-risk ratio evaluation at treatment initiation or follow-up.

   The evaluation of this type of side effect is not easy from a methodological point of view and there are almost no data on this subject except for the most recent antiepileptics. In addition, this type of side effect is not always reported by children. Parents, on the other hand, do not easily notice cognitive effects when starting treatment, whereas they observe a difference when stopping the drug.The cognitive domains where antiepileptics have been shown to have a negative effect are speed of treatment and attention processes. Reviews of the cognitive effects of antiepileptics do not focus on benzodiazepines and there are no data on the cognitive effect of benzodiazepines on children in the general population to our knowledge. This may be because there are not only very few controlled or open studies that have sought to assess the cognitive effects of benzodiazepines used as a treatment in children with epilepsy. Clobazam appears to have like the other antiepileptic drugs some cognitive side effect. A number of studies that have been conducted in children with active epilepsy or epileptic encephalopathy suggest that the use of a benzodiazepine as an anti-epileptic treatment has a positive effect. This may be explained by the suppression of seizures or the suppression of the epileptic encephalopathy process, which have a greater cognitive effect than drugs. More recently, the study by Boshusein et al. used an interesting methodology that, once modified, would make it possible to assess the cognitive role of antiepileptics and to avoid the consequences of repeated seizures. These authors investigated the cognitive effect of discontinuation of treatment by comparing data from an intelligence quotient test (IQ) before and after epilepsy surgery showing that discontinuation of treatment (and cessation of seizures through surgery) was responsible for an increase in IQ.
4. Benefits and risks for research participants It is difficult to assess the impact of antiepileptic drugs in children with epilepsy because the effect of treatments cannot be distinguished from the impact of repeated seizures. The originality here is our methodology which will allow us to have an analysis of the impact of the drug alone.

   The investigators will conduct a prospective study on the cognitive impact of benzodiazepine withdrawal after epilepsy control after epilepsy surgery in children.

   The investigators will focus, through neuropsychological tests, on the working memory and attention abilities of children with drug-resistant epilepsy who require surgery and are receiving a benzodiazepine. The three assessments (pre-surgical (seizures and benzodiazepine); post-surgical (no seizure and benzodiazepine) and after benzodiazepine discontinuation (no seizure and benzodiazepine) will assess the impact of benzodiazepines on working memory and attention span.
5. Objectives Main objective: The main objective is to evaluate the impact on working memory of benzodiazepine discontinuation in children after epilepsy surgery.

   Secondary objectives: Evaluate the impact of benzodiazepine discontinuation on these same children on:

   Short-term memory and visuospatial memory Attention in its different forms Attention and speed of the visual attention Attention and speed on the sensorimotor level Attention and speed at the executive level
6. Description of the research methodology Experimental design: This is a prospective cohort study, in which patients who will be operated on for respective epilepsy surgery in the case of focal epilepsy

This study will include 3 visits:

1. The first visit (V1) will allow for inclusion and first cognitive assessment, before surgery and with benzodiazepines. The purpose of this visit is to include the patient and the first cognitive assessment that will reflect the impairment associated with epilepsy with repeated seizures. At most, a delay of 3 months will occur between the V1 visit and surgery, although in healthcare practice is often shorter.
2. The second visit will take place 3 months after the surgery without any modification of the treatments (V2). It will allow for clinical reassessment (healing or presence seizure) as well as a new cognitive assessment, after surgery and with benzodiazepines. This visit will reflect the cognitive functioning after the surgical procedure. This visit will allow to evaluate the epilepsy status of the child after surgery. The decrease in benzodiazepine will be initiated from V2 over 3 to 6 months depending on the choice of the prescriber, as is usually done in practice. This decrease will be achieved as part of the care, and offered to children who have been seizure free for at least 1 month at the time of V2.
3. The third visit will allow the collection of clinical data and a new cognitive evaluation, after surgery and 3 months after the complete discontinuation of benzodiazepine (V3). This visit will provide data reflecting the cognitive consequences of the benzodiazepines withdraw. The decrease in benzodiazepine will be initiated from V2 over 3 to 6 months depending on the choice of the prescriber, as is usually done in practice. Visit 3 will therefore be between 9 and 12 months after the surgery. It is possible in rare cases that complete discontinuation of benzodiazepine may not be possible, in which case the assessment will be made 3 months after a stable and lower dose of benzodiazepine.

   * It is therefore the evolution of cognitive functions between V2 and V3 that will make possible to meet the main objective. Visit 1 will allow the selection of the patient, it will also allow to have an assessment in comparison with V2 to evaluate the cognitive impact of the surgery combined with the presence or absence of repeated seizures according to each patient.
   * There is no control group planned in this study. The investigators do not expect any change in cognitive functions of children with epilepsy if no major modification of treatment
   * From a regulatory point of view, this is biomedical research, but only neuropsychological assessments are carried out as a result of the research. All other diagnostic and therapeutic actions (and in particular surgery and epilepsy and the reduction of antiepileptic treatment) are performed as part of the care

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria :
* Children aged 6 years to 14 years and 10 months
* Epilepsy patients with drug-resistant focal epilepsy with programmed curative surgical management
* Subject with IQ greater than 70 (Evaluation of IQ in pre-surgical evaluation)
* Antiepileptic drug regimen comprising a benzodiazepine daily
* Subject beneficiary of French national social security scheme
* Parental (and the child if he or she is of age to do so) have signed the study consent

Exclusion Criteria:

* Patient unable to perform cognitive tests or unwilling to do them
* Planned change in drug regimen before the post-surgical period
* Denied to participate in the research

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients will be included among children being followed for drug-resistant epilepsy in pre-surgical assessment by the coordinator team or one of the partners.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Working memory (Digits Backward - Digit Span assessment) from Visit 2 to visit 3 (aka before and after benzodiazepine discontinuation) in post surgical seizure free children | Two assessments will be conducted: One in post-operative seizure-free patient at 3-month postoperative visit (visit 2, before benzodiazepine tapering) and a second at 3-month visit after benzodiazepine discontinuation (visit 3)
  For this test (Digit Span assessment), the examiner tells the child a series of increasingly long numbers and asks the child to repeat this series of numbers from the last to the first. This is a standardized (age-specific) test with a score from 1 to 19 with an average score of 10. This test is used to evaluate the working memory.

SECONDARY OUTCOMES:
Change in short-term memory (Digits Forward - Digit Span assessment) from before to after benzodiazepine discontinuation in post surgical seizure free children | Two assessments will be conducted: One in post-operative seizure-free patient at 3-month postoperative visit and a second at 3-month visit after benzodiazepine discontinuation
  The examiner tells the child a series of increasingly long numbers that he must repeat immediately after the examiner in the same order as the one presented (2 numbers, then 3 numbers,...). This is a standardized (age-specific) test with a score from 1 to 19 with an average score of 10. This test is used to evaluate short-term memory
Change in spacial working memory (forward Corsi Block) from before to after benzodiazepine discontinuation in post surgical seizure free children | Two assessments will be conducted: One in post-operative seizure-free patient at 3-month postoperative visit and a second at 3-month visit after benzodiazepine discontinuation
  The examiner presents a board to the child on which are glued small identical cubes. The examiner will touch 2 cubes successively with the index finger and asks the child to touch the same cubes in the same order as him, then 3 cubes, then 4 cubes,... This is a standardized test (on age). This test is used to evaluate visuo-spacial short-term memory
Change in spacial working memory (backward Corsi Block) from before to after benzodiazepine discontinuation in post surgical seizure free children | Two assessments will be conducted: One in post-operative seizure-free patient at 3-month postoperative visit and a second at 3-month visit after benzodiazepine discontinuation
  The examiner presents a board to the child on which are glued small identical cubes. The examiner will touch with the index finger successively 2 cubes (then 3 cubes,...) and asks the child to touch the cubes starting with the last one until the 1st. This is an age-standardized test. This test is used to evaluate the spacial working memory
Change in attention (TEA-Ch ("Test of Everyday Attention for Children")) from before to after benzodiazepine discontinuation in post surgical seizure free children | Two assessments will be conducted: One in post-operative seizure-free patient at 3-month postoperative visit and a second at 3-month visit after benzodiazepine discontinuation
  This standardized test is used to evaluate the different components of attention. This is a test commonly used to study attention functions from 1h30 to 2h. TEA-Ch makes it possible to establish a diagnosis of attention deficit but above all to define more precisely the deficient modality: sustained attention, focused attention and attentional control. Different tests are proposed (search in the sky, gunfire, do two things at a time, listen to two things at a time...). There are two forms A and B that test the effect of an intervention to modify attention (to avoid the retest effect). This is a standardized test (on age).
Change in visual attention and visual rapidity from before to after benzodiazepine discontinuation in post surgical seizure free children benzodiazepine discontinuation in post surgical seizure free children | Two assessments will be conducted: One in post-operative seizure-free patient at 3-month postoperative visit and a second at 3-month visit after benzodiazepine discontinuation
  This is a 1-minute timed target barrage test (rabbits and cats for the youngest and female and male faces for the oldest). It is a A Developmental Neuropsychological Assessment(NEPSY) subtest. It is a question of discriminating against one of the two entities. The number of targets analyzed by the patient allows us to score the level of attention. This is a standardized test (on age).
Change in executive function attention and rapidity (Purdue Pegboard test) from before to after benzodiazepine discontinuation in post surgical seizure free children | Two assessments will be conducted: One in post-operative seizure-free patient at 3-month postoperative visit and a second at 3-month visit after benzodiazepine discontinuation
  This is a timed test where the child must place rods in holes for 1 minute: first with the dominant hand, then the non-dominant hand and then in a two-handed situation. This is a standardized test (on age).

CONTACTS AND LOCATIONS:
Overall Officials: Adina ILEA, Dr, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Robert-Debré, Paris, Île-de-France Region, France